CLINICAL TRIAL: NCT04326309
Title: Audio Data Collection for Identification and Classification of Coughing
Status: Completed | Type: Observational
Sponsor: HealthMode Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM070102
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Coronavirus Infections; Hay Fever; Asthma; Chronic Obstructive Pulmonary Disease; Influenza; Common Cold; Respiratory Tract Infections; Healthy
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Rhinitis, Allergic, Seasonal; Asthma; Pulmonary Disease, Chronic Obstructive; Influenza, Human; Common Cold; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Individual Application Downloaders
- Cohort 2: Public Space and Vehicle Data Capture
- Cohort 3: Individuals dialing a voice-recording study phone number
- Cohort 4: Individuals utilizing study website's audio recording functionality
- Cohort 5: Individuals participating in Return-to-Work Project

SUMMARY:
An open access study that will define and collect digital measures of coughing in multiple populations and public spaces using various means of audio data collection.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1, 3, 4 and 5:

* Females and males over 18 years old
* Willing to share demographic data with the sponsor of the study
* Willing to follow app use instructions during the course of the study
* Willing to complete survey instruments as described in study procedures
* Willing to provide electronic informed consent
* Able to read and understand the English language well enough to complete electronic informed consent

Cohort 2:

Any person present in the vicinity of a HealthMode Cough Monitoring Device

Exclusion Criteria:

No exclusion criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US resident participants downloading the HealthMode Stool application from the Apple AppStore (Cohort 1) and persons in the vicinity of a HealthMode Cough Monitoring Device (Cohort 2)
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Dataset size | 14 days
  Size of collected audio dataset measured as number of collected cough sounds, targeting ≥10,000 identified coughs.

SECONDARY OUTCOMES:
Cough sound identification | 14 days
  Identification of cough sounds by the existing mathematical model with ≥ 99% specificity and ≥ 60% sensitivity
Improvement of the existing model | 14 days
  Increase in the sensitivity of the mathematical model to cough sounds to ≥ 70% while retaining the specificity of ≥ 99%
Evaluate the usability of the application | 14 days
  Determination of the level of acceptance and satisfaction of the solution by patients by means of a Standard Usability Questionnaire to provide feedback. The score ranges from 10 to 50, higher score indicating a better usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual Facility, The Bronx, New York, United States